CLINICAL TRIAL: NCT00108407
Title: Integrated CBT for Substance Use and Depressive Disorders
Brief Title: Study Comparing Two Types of Psychotherapy for Treating Depression and Substance Abuse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Brown, Sandra - Principal Investigator, Department of Veterans Affairs
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: MHBS-041-99Sa
Record Dates: First submitted 2005-04-14; First posted 2005-04-15 (Estimated); Last update posted 2009-03-06 (Estimated); Status verified 2009-03

CONDITIONS: Alcohol Abuse; Cannabis Abuse; Major Depressive Disorder; Substance-Related Disorders
Keywords: Alcohol Abuse/Dependence; Alcohol Use Disorders; Cannabis Abuse/Dependence; Depression; Dual diagnosis; Dysthymia; Stimulant Abuse/Dependence; Substance Use Disorders
MeSH Terms: conditions — Alcoholism; Marijuana Abuse; Depressive Disorder, Major; Substance-Related Disorders; Depression; Dysthymic Disorder

ARMS (2):
- 1 (Experimental): Integrated Cognitive Behavioral Therapy
  Interventions: Behavioral: Integrated Cognitive Behavioral Therapy
- 2 (Experimental): Twelve Step Facilitation Therapy
  Interventions: Behavioral: Twelve Step Facilitation Therapy

INTERVENTIONS:
Behavioral: Integrated Cognitive Behavioral Therapy
  Arms: 1
Behavioral: Twelve Step Facilitation Therapy
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether Integrated Cognitive Behavioral Therapy or Twelve Step Facilitation Therapy is most effective for treatment of dually diagnosed veterans with depressive and substance use disorders.

DETAILED DESCRIPTION:
Depression is the most frequent co-occuring mental health disorder among adults with substance use disorders, and such comorbidity is often associated with poorer treatment outcomes. Although there is an urgent need for effective treatments specific for dual-diagnosis adults, few studies have been conducted to address this need.

Comparison: This study will compare substance use and depression symptoms of individuals in two different psychotherapy groups: Integrated Cognitive Behavioral Therapy and Twelve Step Facilitation Therapy. Symptoms and substance use will be compared during the active treatment phase (24 weeks) and for one year following the end of the active treatment.

ELIGIBILITY:
Inclusion Criteria:

* Individuals diagnosed with one or more substance use disorders (alcohol, cannabis, and or stimulant abuse/dependence) and an independent co-occurring depressive disorder (major depression or dysthymia) will be included.

Exclusion Criteria:

* Individuals with substance induced mood disorders and individuals experiencing persistent psychotic symptoms.
* Those with life threatening or unstable medical illness, neurological disorders, or inability to read will be excluded.
* Individuals currently prescribed steroids, disulfiram, or long acting benzodiazepines will be excluded.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-10

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Brown, PhD, Principal Investigator — VA San Diego Healthcare System, San Diego
Locations (1):
- VA San Diego Healthcare System, San Diego, San Diego, California, United States

REFERENCES:
- [Derived] Worley MJ, Tate SR, Granholm E, Brown SA. Mediated and moderated effects of neurocognitive impairment on outcomes of treatment for substance dependence and major depression. J Consult Clin Psychol. 2014 Jun;82(3):418-28. doi: 10.1037/a0036033. Epub 2014 Mar 3. PMID 24588403
- [Derived] Tripp JC, Skidmore JR, Cui R, Tate SR. Impact of Physical Health on Treatment for Co-occurring Depression and Substance Dependence. J Dual Diagn. 2013;9(3):10.1080/15504263.2013.806111. doi: 10.1080/15504263.2013.806111. PMID 24223036
- [Derived] Worley MJ, Tate SR, McQuaid JR, Granholm EL, Brown SA. 12-step affiliation and attendance following treatment for comorbid substance dependence and depression: a latent growth curve mediation model. Subst Abus. 2013;34(1):43-50. doi: 10.1080/08897077.2012.691451. PMID 23327503
- [Derived] Worley MJ, Tate SR, Brown SA. Mediational relations between 12-Step attendance, depression and substance use in patients with comorbid substance dependence and major depression. Addiction. 2012 Nov;107(11):1974-83. doi: 10.1111/j.1360-0443.2012.03943.x. Epub 2012 Aug 10. PMID 22578037